CLINICAL TRIAL: NCT05143788
Title: Strategic Intervention on Preserving Motor Function With Application of Monopolar Stimulator During Awake Glioma Resection Surgery
Brief Title: Strategic Intervention on Preserving Motor Function During Awake Craniotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Neurosurgical Institute (Other)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JYY-2019-5
Record Dates: First submitted 2021-11-23; First posted 2021-12-03 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-11

CONDITIONS: Glioma
Keywords: glioma; awake craniotomy; motor function; recovery
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New surgical plan group (Experimental): The investigators use monopolar stimulators to determine and retain the tumor margin within 5mm from the posterior limb of the inner capsule in type III motor area glioma patients.
  Interventions: Procedure: Awake craniotomy
- Traditional surgical plan group (Active Comparator): The investigators use bipolar stimulator according to the current standard surgery plan. After the positive points are identified by stimulator, the positive points are retained in order to preserve the motor function while all the non-positive points of the tumor are resected.
  Interventions: Procedure: Awake craniotomy

INTERVENTIONS:
Procedure: Awake craniotomy — The awake neurosurgical procedure performed on the brain is to provide a real-time neurological functions monitoring in order to preserve the functions of brain to the greatest extent.

SUMMARY:
This study aims to compare the motor functions after traditional or a new surgical plan during awake glioma resection surgery.

DETAILED DESCRIPTION:
This study concentrates on patients with type III motor area glioma. In the awake surgery, The investigators compare the new surgical plan, which the investigators use a monopolar stimulator to determine and retain the tumor margin within 5mm from the posterior limb of the inner capsule. For the traditional surgical plan, the investigators use bipolar stimulator according to the current standard surgery plan. After the positive points are identified by stimulator, the positive points are retained in order to preserve the motor function while all the non-positive points of the tumor are resected. This study is designed to determine whether the new surgical plan is more suitable for type III motor area glioma patients.

ELIGIBILITY:
Inclusion Criteria:

* 1)Age ≥ 18 years <65 years; 2)Histopathological diagnosis with low grade glioma (LGG) according to the 2021 World Health Organization (WHO) criteria; 3)Patients with primary type III (the tumor is less than 5 mm away from the posterior limb of the inner capsule) supratentorial glioma in the motor area confirmed by radiologist; 4)No history of biopsy, radiotherapy, or chemotherapy.

Exclusion Criteria:

* 1) Patients who received radiotherapy, chemotherapy or anti-tumor biotherapy within 1 month before the test; 2) Patients who received immunotherapy within 3 months before the test; 3) Patients who participated in other clinical trials within 3 months before the test ; 4) Patients with a history of severe allergies or allergies; 5) Pregnancy, breastfeeding or those who are fertile but have not taken contraceptive measures; 6) Have other serious medical diseases or severe uncontrollable infections; 7) Drugs and drugs Abuse, long-term alcoholism and AIDS patients; 8) Those who have uncontrollable seizures, or lose self-control due to mental illness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Motor function preserved better in new surgical plan group | through study completion, an average of 2 years
  Motor function of the participants in new surgical plan group is better preserved and recover faster than the participants in traditional surgical group.The difference between the motor functions of two groups are analyzed using t-test or chi-square test according to the type of data.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Jiang, MD and PhD, Study Director — Beijing Neurosurgical Institute and Beijing Tiantan Hospital

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share individual participant data with other researchers

REFERENCES:
- [Result] Fang S, Li Y, Wang Y, Zhang Z, Jiang T. Awake craniotomy for gliomas involving motor-related areas: classification and function recovery. J Neurooncol. 2020 Jun;148(2):317-325. doi: 10.1007/s11060-020-03520-w. Epub 2020 Apr 29. PMID 32350781